CLINICAL TRIAL: NCT02337829
Title: A Phase II Study Using ACP-196 (Acalabrutinib) in Patients With Relapsed/Refractory and Treatment-naïve Deletion 17p CLL/SLL: Pharmacodynamic Assessment of BTK Inhibition and Antitumor Response.
Brief Title: Acalabrutinib in Patients With Relapsed/Refractory and Treatment naïve Deletion 17p CLL/SLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-H-0016
Record Dates: First submitted 2014-11-19; First posted 2015-01-14 (Estimated); Results first posted 2021-08-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Relapsed/refractory CLL; Btk; Leukemia; Lymphocytic; Lymphoma; Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); ACP-196; Acalabrutinib; Treatment naive CLL; 17p deletion; TP53 mutation; NOTCH1 mutation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia; Lymphoma; Chromosome 17 deletion | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Subjects will be randomized to receive 1 of 2 dosing regimens: 1) acalabrutinib, dose A once daily; or 2) acalabrutinib, dose B twice daily.
  Interventions: Drug: Acalabrutinib (Arm A); Drug: Acalabrutinib (Arm B)
- Arm B (Experimental): Subjects will be randomized to receive 1 of 2 dosing regimens: 1) acalabrutinib, dose A once daily; or 2) acalabrutinib, dose B twice daily.
  Interventions: Drug: Acalabrutinib (Arm A); Drug: Acalabrutinib (Arm B)

INTERVENTIONS:
Drug: Acalabrutinib (Arm A) — * A1a) acalabrutinib, dose A daily: biopsy (T) schedule W;
  * A1b) acalabrutinib, dose A daily: biopsy (T) schedule V.
  * A2a) acalabrutinib, dose B q 12 hours: biopsy (T) schedule Y;
  * A2b) acalabrutinib, dose B q 12 hours; biopsy (T) schedule Z
  Other Names: ACP-196
Drug: Acalabrutinib (Arm B) — B1c) acalabrutinib, dose A daily: biopsy (U) schedule W;
  • B2c) acalabrutinib, dose B q12 hours: biopsy (U)) schedule Y.
  Other Names: ACP-196

SUMMARY:
This study is to determine the response to acalabrutinib in patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
To investigate the safety and efficacy of acalabrutinib for patients with CLL/SLL that have relapsed/refractory disease or treatment naive deletion 17p.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older with histologically confirmed disease.
* Active disease as defined by at least one of the following (IWCLL consensus criteria):

  * Weight loss ≥10% within the previous 6 months
  * Extreme fatigue
  * Fevers of greater than 100.5ºF for ≥2 weeks without evidence of infection
  * Night sweats for more than one month without evidence of infection
  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
  * Massive or progressive splenomegaly
  * Massive nodes or clusters or progressive lymphadenopathy
  * Progressive lymphocytosis with an increase of >50% over a 2 month period, or an anticipated doubling time of less than 6 months
  * Compensated autoimmune hemolysis
* Relapsed/Refractory CLL or treatment naïve CLL patients with 17p deletion, TP53 mutation, or NOTCH1 mutation
* Agreement to use acceptable methods of contraception during the study and for 30 days after the last dose of study drug if sexually active and able to bear or beget children.
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty and serial biopsies.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Exclusion Criteria:

* Radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or investigational products in the last 4 weeks.
* Richter's transformation. Autoimmune hemolytic anemia or thrombocytopenia requiring steroid therapy. Impaired hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2025-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Clinical Study Information Center, Study Director — 1-877-240-9479 - information.center@astrazeneca.com
Locations (1):
- Research Site, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Alsadhan A, Chen J, Gaglione EM, Underbayev C, Tuma PL, Tian X, Freeman LA, Baskar S, Nierman P, Soto S, Itsara A, Ahn IE, Sun C, Bibikova E, Hartmann TN, Mhibik M, Wiestner A. CD49d Expression Identifies a Biologically Distinct Subtype of Chronic Lymphocytic Leukemia with Inferior Progression-Free Survival on BTK Inhibitor Therapy. Clin Cancer Res. 2023 Sep 15;29(18):3612-3621. doi: 10.1158/1078-0432.CCR-22-3217. PMID 37227160
- [Derived] Cyr MG, Mhibik M, Qi J, Peng H, Chang J, Gaglione EM, Eik D, Herrick J, Venables T, Novick SJ, Courouble VV, Griffin PR, Wiestner A, Rader C. Patient-derived Siglec-6-targeting antibodies engineered for T-cell recruitment have potential therapeutic utility in chronic lymphocytic leukemia. J Immunother Cancer. 2022 Nov;10(11):e004850. doi: 10.1136/jitc-2022-004850. PMID 36442911
- [Derived] Sun C, Nierman P, Kendall EK, Cheung J, Gulrajani M, Herman SEM, Pleyer C, Ahn IE, Stetler-Stevenson M, Yuan CM, Maric I, Gaglione EM, Harris HM, Pittaluga S, Wang MH, Patel P, Farooqui MZH, Izumi R, Hamdy A, Covey T, Wiestner A. Clinical and biological implications of target occupancy in CLL treated with the BTK inhibitor acalabrutinib. Blood. 2020 Jul 2;136(1):93-105. doi: 10.1182/blood.2019003715. PMID 32202637
- [Derived] Alsadhan A, Cheung J, Gulrajani M, Gaglione EM, Nierman P, Hamdy A, Izumi R, Bibikova E, Patel P, Sun C, Covey T, Herman SEM, Wiestner A. Pharmacodynamic Analysis of BTK Inhibition in Patients with Chronic Lymphocytic Leukemia Treated with Acalabrutinib. Clin Cancer Res. 2020 Jun 15;26(12):2800-2809. doi: 10.1158/1078-0432.CCR-19-3505. Epub 2020 Feb 13. PMID 32054731
- See also: 15-H-0016_Protocol Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15-H-0016&attachmentIdentifier=e4575fcb-4235-4e46-a0ef-ba83d6d840e2&fileName=15-H-0016-protocol_Redacted.pdf&versionIdentifier=
- See also: 15-H-0016_SAP ed.3 Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15-H-0016&attachmentIdentifier=c6643522-782d-4db3-8af9-8823ea068dc4&fileName=15-h-0016-sap-ed-3_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Acalabrutinib 100 mg BID Relapse/Refractory: relapsed/refractory subjects treated with acalabrutinib 100 mg twice a day
- Acalabrutinib 200 mg QD Relapse/Refractory: Relapse/Refractory subjects treated with acalabrutinib 200 mg once a day
- Acalabrutinib 100 mg BID Treatment Naive: Treatment naive subjects treated with acalabrutinib 100 mg twice a day
- Acalabrutinib 200 mg QD Treatment Naive: Treatment naive subjects treated with acalabrutinib 200 mg once a day
Period: Overall Study
Arm/Group | Acalabrutinib 100 mg BID Relapse/Refractory | Acalabrutinib 200 mg QD Relapse/Refractory | Acalabrutinib 100 mg BID Treatment Naive | Acalabrutinib 200 mg QD Treatment Naive
Started | 18 | 14 | 6 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 18 | 14 | 6 | 10
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 12 | 10 | 5 | 6
Not completed — discontinued for other reasons | 6 | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acalabrutinib 100 mg BID Relapse/Refractory | Acalabrutinib 200 mg QD Relapse/Refractory | Acalabrutinib 100 mg BID Treatment Naive | Acalabrutinib 200 mg QD Treatment Naive | Total
Number analyzed (Participants) | 18 | 14 | 6 | 10 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (9.3) | 62.3 (7.7) | 68.3 (10.9) | 62.1 (8.7) | 63.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 2 | 4 | 15
  Male | 12 | 11 | 4 | 6 | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 14 | 6 | 9 | 47
  Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 2
  Black or African American | 2 | 0 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 16 | 12 | 4 | 7 | 39
  Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: Participants]
  United States | 18 | 14 | 6 | 10 | 48

OUTCOME MEASURES:

1. Primary Outcome: Response Based on Overall Response Rate
Description: The best response to treatment was determined according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria incorporating 2012 and 2013 clarifications pertaining to subjects treated with kinase inhibitors. Overall response rate (ORR) was the proportion of subjects who achieved complete response (CR), CR with incomplete marrow recovery (CRi), or partial response (PR) while on treatment before the initiation of new anti-cancer therapy or stem cell transplant.
Time Frame: Cycle 1 (28 Days) to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Total Relapse/Refractory Subjects: All relapse/refractory subjects in both dose groups combined
- Total Treatment Naive Subjects: All treatment naive subjects in both dose groups combined
Arm/Group | Acalabrutinib 100 mg BID Relapse/Refractory | Acalabrutinib 200 mg QD Relapse/Refractory | Total Relapse/Refractory Subjects | Acalabrutinib 100 mg BID Treatment Naive | Acalabrutinib 200 mg QD Treatment Naive | Total Treatment Naive Subjects
Number analyzed (Participants) | 18 | 13 | 31 | 6 | 10 | 16
Participants | 17 | 11 | 28 | 6 | 8 | 14

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days post last dose for each subject; an average of approximately 38 months.
Arm/Group | Acalabrutinib 100 mg BID Relapse/Refractory | Acalabrutinib 200 mg QD Relapse/Refractory | Acalabrutinib 100 mg BID Treatment Naive | Acalabrutinib 200 mg QD Treatment Naive
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/14 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 11/18 | 8/14 | 3/6 | 5/10
Other Adverse Events (participants affected / at risk) | 18/18 | 14/14 | 6/6 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib 100 mg BID Relapse/Refractory (N=18) | Acalabrutinib 200 mg QD Relapse/Refractory (N=14) | Acalabrutinib 100 mg BID Treatment Naive (N=6) | Acalabrutinib 200 mg QD Treatment Naive (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatitis b reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib 100 mg BID Relapse/Refractory (N=18) | Acalabrutinib 200 mg QD Relapse/Refractory (N=14) | Acalabrutinib 100 mg BID Treatment Naive (N=6) | Acalabrutinib 200 mg QD Treatment Naive (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglobulinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (3) | 3 (3) | 1 (1) | 2 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lenticular opacities (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (2) | 0 (0) | 1 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (12) | 7 (13) | 4 (5) | 4 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8) | 6 (7) | 2 (2) | 3 (7)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Poor dental condition (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6) | 0 (0) | 2 (4)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 5 (6) | 4 (6) | 3 (4)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 7 (14) | 9 (15) | 3 (6) | 8 (15)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 3 (3) | 1 (3) | 0 (0) | 3 (4)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 4 (5) | 5 (7) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (2) | 2 (3) | 2 (2)
Pyrexia (General disorders) | 4 (5) | 3 (3) | 0 (0) | 4 (9)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 2 (3) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema migrans (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Lip infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (4) | 1 (1) | 3 (3)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (8) | 3 (3) | 3 (4) | 1 (1)
Skin infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (13) | 6 (12) | 3 (4) | 5 (10)
Urinary tract infection (Infections and infestations) | 3 (7) | 3 (3) | 2 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 1 (1) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 11 (16) | 9 (14) | 6 (11) | 6 (12)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Beta 2 microglobulin increased (Investigations) | 2 (2) | 1 (3) | 1 (3) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 3 (5) | 2 (2) | 0 (0) | 4 (7)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood urea decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Cd4 lymphocytes decreased (Investigations) | 6 (7) | 4 (8) | 3 (4) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (8) | 3 (13) | 3 (10) | 0 (0)
Lymphocyte count increased (Investigations) | 3 (4) | 3 (3) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (6) | 6 (11) | 1 (1) | 1 (5)
Neutrophil count increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 4 (14) | 2 (2) | 2 (7) | 3 (5)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (4) | 4 (9) | 1 (2) | 2 (2)
Weight increased (Investigations) | 5 (13) | 3 (9) | 4 (12) | 2 (4)
White blood cell count decreased (Investigations) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (10) | 4 (8) | 3 (5) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (8) | 3 (7) | 5 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (3) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 8 (13) | 1 (2) | 5 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 5 (6) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (7) | 5 (5) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 12 (20) | 10 (15) | 5 (10) | 6 (11)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (5) | 0 (0) | 2 (3)
Phonophobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (5) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (4) | 2 (2) | 3 (3) | 1 (2)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrometra (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 2 (2) | 3 (4) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7) | 3 (5) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (3) | 0 (0) | 1 (3)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 3 (3) | 2 (2) | 4 (4)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (4) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (4)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5) | 0 (0) | 5 (8)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7) | 8 (17) | 1 (1) | 4 (6)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibromuscular dysplasia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 2 (2) | 1 (2) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 10 (32) | 7 (13) | 3 (8) | 2 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT02337829/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT02337829/SAP_004.pdf